CLINICAL TRIAL: NCT04889963
Title: Regeneration of Posterior Cruciate Ligament Injury Using Hypoxia Conditioned Allogenic Adipose Mesenchymal Stem Cell (AdMSC) and Ligament Derived Condition Medium (Secretome)
Brief Title: Regeneration of Posterior Cruciate Ligament Injury Using Hypoxic Conditioned Allogenic Adipose Mesenchymal Stem Cell and Condition Medium
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Sholahuddin Rhatomy, Director, Head of Orthopaedic Department,faculty of medicine,public health and nursing,universitas gadjah mada, Sholahuddin Rhatomy,MD, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STEMCELL-LIGAMENTREGENERATION
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Adypose Mesenchimal Stem Cell; Ligament Rupture; Ligament Derived Conditined Medium
Keywords: adypose mesenchimal stem cell hypoxic culture conditioned; Ligament Rupture; ligament derived conditined medium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Placebo Comparator): rabbit with posterior cruciate ligament rupture and treated with fibrin glue (sacffold)
  Interventions: Biological: adypose mesenchymal conditioned medium and ligament derived conditioned medium
- conditioned medium group (Active Comparator): rabbit with posterior cruciate ligament rupture and treated with fibrin glue mix with ligament derived conditioned medium
  Interventions: Biological: adypose mesenchymal conditioned medium and ligament derived conditioned medium
- stem cells group (Active Comparator): rabbit with posterior cruciate ligament rupture and treated with fibrin glue mix with adypose mesenchymal stem cells in hypoxic culture condition
  Interventions: Biological: adypose mesenchymal conditioned medium and ligament derived conditioned medium
- composite group (Experimental): rabbit with posterior cruciate ligament rupture and treated with fibrin glue mix with adypose mesenchymal stem cells in hypoxic culture condition and ligament derived conditioned medium
  Interventions: Biological: adypose mesenchymal conditioned medium and ligament derived conditioned medium

INTERVENTIONS:
Biological: adypose mesenchymal conditioned medium and ligament derived conditioned medium — rabbit with posterior cruciate ligament rupture and treated with fibrin glue mix with adypose mesenchymal stem cells in hypoxic culture and ligament derived conditioned medium

SUMMARY:
Transplantation of Allogenic Adipose Mesenchimal Stem cell in hypoxic cultur condition with Ligament- derived conitioned medium can enhance regeneration of posterior cruciate ligament rupture

DETAILED DESCRIPTION:
this study is in vivo study to prove effect of transplantation of Allogenic Adipose Mesenchimal Stem cell in hypoxic cultur condition with Ligament- derived conitioned medium in regeneration of posterior cruciate ligament rupture

ELIGIBILITY:
Inclusion Criteria:

* white male new zealand rabbit
* weight 2500 - 3000 gram

Exclusion Criteria:

* have no disease

Ages: 2 Months to 12 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — white male rabbit
Enrollment: 16 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
tensile strength of posterior cruciate ligament | 6 weeks
  measurement of tensile strength of posterior cruciate ligament
Thrombosite of Growth Factor - beta 1 | 6 weeks
  measurement value of Thrombosite Growth Factor - beta 1
basic fibroblast of growth factor | 6 weeks
  measurement value of basic fibroblast of growth factor

CONTACTS AND LOCATIONS:
Locations (1):
- Sholahuddin Rhatomy, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided